CLINICAL TRIAL: NCT00115401
Title: Gait Adaptations to Passive Dynamic Ankle-Foot Orthosis Use
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050175; 05-CC-0175
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-17

CONDITIONS: Joint Instability
Keywords: Walking; Compensation; Leg Weakness; Orthotics; Joint Impairment; Healthy Volunteer; HV; Joint Inmpairment
MeSH Terms: conditions — Joint Instability

SUMMARY:
This study will collect information on the different ways that people walk, that is, their gait, when they use ankle braces. Patients will visit NIH on at least three and as many as nine separate occasions. A physical therapist will perform a physical examination to determine how patients move, how strong they are and what their comfortable walking speed is. Then patients will sit on a chair while a camera apparatus takes special pictures of their legs, a procedure lasting up to 2 hours. Patients will be asked to return to learn how to walk with the custom Passive Dynamic Ankle-Foot Orthosis (PD-AFO)-a unique ankle brace designed to improve walking ability by providing natural support to the lower limb.

Patients 4 and older who are in good health and able to walk repeatedly a distance of 15 meters (approximately 49 feet) independently and unsupervised may be eligible for this study.

With this training, patients may return several times to learn how to walk with the brace, but for their protection, they will not be allowed to take it or use it outside the research team's supervision. The researchers will examine the leg to ensure that the brace fits and will ask questions about it. Each training visit will require up to 1.5 hours. When patients have learned to walk with the brace, they will be asked to visit again and walk while scientific pictures are taken of their legs. During the walking test, patients will wear T-shirts and shorts. Patients' arms and legs will be wrapped with a soft, rubber-like material, to allow small plastic reflective balls to be attached. Firm material known as a shell can be attached to the rubber sleeves, with Velcro or a self-sticking bandage. The small balls may also be attached to the skin, with an adhesive. Also, there may be a test of the muscles, through the use of electromyography, or EMG. The test involves attachment of small metal electrodes to the surface of the skin, again with an adhesive. There should not be discomfort with that test.

As patients walk several times, scientific cameras will record the positions of the reflective balls. Pictures do not involve patients' faces or other parts of the body. Afterward, a unique chair system called a Biodex will measure the leg muscle strength. Patients will be asked to sit on the chair and place their leg in a foot in an apparatus, a special structure that measures strength. They will repeatedly push against the apparatus, doing so for 3 seconds. Each time patients push, the researchers will touch a small magnetic device to the skin, which will cause the muscles to push harder. Although this procedure should not cause any discomfort, it may feel unusual. If they wish, patients can ask to stop the test at any time. Few risks are involved in participating in this series of activities. There is a slight chance of mild skin irritation from the adhesives used on the skin or from the soft, rubber-like material. But the material is worn for only a brief period, and skin reactions are rare. Also, that material may feel tight, but if it causes discomfort or prevents moving, patients can ask a researcher to adjust it. There is a slight chance of skin irritation from use of the PD-AFO, but adjustment can be made to make patients comfortable. Patients may experience some muscle soreness caused by participating in the muscle strength tests. However, they will be safely monitored by a physical therapist when they try on the brace to adjust to its feel and fit, as well as during testing of gait.

This study will not have a direct benefit for participants. However, participants will be paid for their time, with minimum compensation of $50.

DETAILED DESCRIPTION:
Ankle-Foot Orthoses are a common form of ankle joint bracing prescribed for patients with impaired joint function. Passive Dynamic Ankle-Foot Orthoses (PD-AFOs) constitute a special class of ankle braces designed to enhance gait function by providing natural support to the lower limb as it progresses over the stance foot. However, a fundamental design characteristic of all PD-AFOs is that they are not capable of replicating all dynamic characteristics of the natural ankle complex. As a result, the efficient use of PD-AFOs during gait requires the wearer to develop an adapted, lower limb movement control strategy that effectively optimizes positive PD-AFO characteristics while compensating for characteristics detrimental to gait function. The long term goal of this research effort is to predict a patient's ability to adapt to PD-AFO use and to customize PD-AFO characteristics to optimize that adaptation. The purpose of this series of studies is to further refine our existing methods of constructing custom PD-AFOs and to document the movement control adaptations produced by normal and healthy strength impaired subjects in response to PD-AFO use.

The research plan is comprised of three phases: technology refinement (pilot) effort (n=5), normal subject study (n=10), and an impaired subject study (n=20). During the technology refinement phase, we will refine our existing methods for PD-AFO customization and pilot test the PD-AFO accommodation gait training methods and movement control assessment measurements. The normal and impaired subject studies will be used to document PD-AFO use under a strength substitution paradigm (normal subject study) and a strength enhancement paradigm (impaired subject study).

Subjects in all study phases will participate in each of three visit types. Initially, subjects will participate in a screening and PD-AFO tuning visit that contains a neuromuscular screening examination, a preferred walking speed test, and measurement for a custom fitting PD-AFO. Following the manufacturing of the custom PD-AFO, subjects will return for their PD-AFO receipt and accommodation training visit. During this visit, the PD-AFO will be further customized and evaluated for comfort and performance and the subject will undergo supervised gait training in PD-AFO use. Following successful accommodation to PD-AFO use, subjects will return for their third visit and undergo instrumented gait analyses under three conditions (targeted walking velocity without the PD-AFO, self selected walking velocity with the PD-AFO, and targeted walking velocity with the PD-AFO) and finally, objective plantarflexor strength testing.

Walking velocity will be statistically compared between with and without PD-AFO conditions to determine the accommodation effect for self selected conditions and to test for differences between targeted walking conditions. The magnitude of peak natural ankle plantarflexion moments will be statistically compared to determine the efficacy of the strength substitution and strength enhancement paradigms. The nature and extent of movement control adaptations will be explored by contrasting the various biomechanical (kinematic and kinetic) variables between with and without PD-AFO conditions having congruent walking speeds. Results of the neurological examination and objective strength testing will be used to rationalize the existence of different movement control adaptations between subjects and form the basis for developing an initial predictive model.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

This study will include healthy males and females who are over four years of age. The study will involve healthy volunteers having normal lower extremity strength profiles and healthy volunteers with impaired ankle joint plantarflexion strength. For this project, the term healthy is defined as a lack of systemic disease that alters ability of subjects to participate in activities of their choice. In addition, healthy means no current pathology where there is any possibility of damage to muscle, ligament, or cartilage in the lower extremity. An attempt will be made to obtain an equal distribution between males and females. In addition, participation of minorities will be strongly encouraged through the use of existing outreach programs.

INCLUSION CRITERIA:

Subjects must be capable of repeatedly walking 15m independently and unsupervised. They must be co-operative and able to follow commands and have adequate natural step and stride lengths to step on three force plates in series. Subjects must have a combined lower limb size (shank and foot) that results in a PD-AFO size within the prototyping capacity (50 cm) of the selective laser sintering machine. To participate in the impaired study, subjects must have a manual muscle strength score for plantarflexion strength that is less than or equal to three out of a five point scale.

EXCLUSION CRITERIA:

Subjects with an unsafe or highly variable gait pattern upon visual observation will be excluded. Subjects who are unable to repeatedly walk through the data collection volume without the use of assistive devices will be excluded. In addition, subjects with pain related to walking or impaired skin sensation (touch and pressure) will be excluded. Subjects with lower extremity muscle spasticity of 3 or greater on the Ashworth Scale will be excluded. Subjects with a history of injury, surgery, or disease affecting the function of the lower extremity will be excluded from the normal study. Subjects will be excluded from participation in the normal study if muscle strength and joint range of motion measures are outside normal limits.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2005-06-16; Study Completion 2007-10-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Holden JP, Chou G, Stanhope SJ. Changes in knee joint function over a wide range of walking speeds. Clin Biomech (Bristol). 1997 Sep;12(6):375-382. doi: 10.1016/s0268-0033(97)00020-x. PMID 11415746